CLINICAL TRIAL: NCT00598975
Title: A Multicenter, Open-Label, Phase 2 Study to Determine the Dose, Safety and Efficacy of NKTR-102 (PEG-Irinotecan) in Combination With Cetuximab in Patients With Solid Tumors Refractory to Standard Treatment and to Evaluate the Safety and Efficacy of NKTR-102 or Irinotecan in Combination With Cetuximab in Second Line, Irinotecan and Cetuximab Naïve, Colorectal Cancer Patients With Metastatic or Locally Advanced Disease
Brief Title: NKTR-102 in Combination With Cetuximab in Patients With Refractory Solid Tumors (Phase 2a) and Metastatic or Locally Advanced Colorectal Cancer (Phase 2b)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-PIR-02
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Tumor; Colorectal Cancer
Keywords: Phase 2a: Multiple solid tumor types; Phase 2b: Second-Line Colorectal Cancer (CRC)
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — etirinotecan pegol; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NKTR-102 100 mg/m2 + Cetuximab (Active Comparator): NKTR-102 100 mg/m2 + Cetuximab Arm
  All patients received NKTR-102 in combination with cetuximab. NKTR-102 was administered intravenously (IV) once every 3 weeks (q3w) over 90 minutes on Day 1. Patients were to be enrolled in one of the following sequential dosing cohorts of NKTR-102: 100, 125, 150, or 175 mg/m2. Only the 100 and 125 mg/m2 were enrolled.
  Interventions: Drug: NKTR-102 100 mg/m2; Drug: Cetuximab
- NKTR-102 125 mg/m2 + Cetuximab (Active Comparator): NKTR-102 125 mg/m2 + Cetuximab Arm
  All patients received NKTR-102 in combination with cetuximab. NKTR-102 was administered intravenously (IV) once every 3 weeks (q3w) over 90 minutes on Day 1. Patients were to be enrolled in one of the following sequential dosing cohorts of NKTR-102: 100, 125, 150, or 175 mg/m2. Only the 100 and 125 mg/m2 were enrolled.
  Interventions: Drug: NKTR-102 125 mg/m2; Drug: Cetuximab

INTERVENTIONS:
Drug: NKTR-102 100 mg/m2 — NKTR-102 100 mg/m2 + Cetuximab Arm:
  All patients received NKTR-102 in combination with cetuximab. NKTR-102 was administered intravenously (IV) once every 3 weeks (q3w) over 90 minutes on Day 1. Patients were to be enrolled in one of the following sequential dosing cohorts of NKTR-102: 100, 125, 150, or 175 mg/m2. Only the 100 and 125 mg/m2 were enrolled.
  Other Names: PEG-Irinotecan
  Arms: NKTR-102 100 mg/m2 + Cetuximab
Drug: NKTR-102 125 mg/m2 — NKTR-102 125 mg/m2 + Cetuximab Arm:
  All patients received NKTR-102 in combination with cetuximab. NKTR-102 was administered intravenously (IV) once every 3 weeks (q3w) over 90 minutes on Day 1. Patients were to be enrolled in one of the following sequential dosing cohorts of NKTR-102: 100, 125, 150, or 175 mg/m2. Only the 100 and 125 mg/m2 were enrolled.
  Other Names: PEG-Irinotecan
  Arms: NKTR-102 125 mg/m2 + Cetuximab
Drug: Cetuximab — Cetuximab was administered once weekly via a 2-hour IV infusion at a starting dose of 400 mg/m2 on Day 1 and subsequently administered weekly at 250 mg/m2 via a 1-hour infusion thereafter.
  Other Names: Erbitux

SUMMARY:
Study 07-PIR-02 is a Phase 2 study designed to evaluate the safety and efficacy of NKTR-102 (PEG-irinotecan) for the treatment of patients with colorectal cancer (CRC). The study is comprised of two sequential components - Phase 2a and Phase 2b. The Phase 2a portion is an open-label, dose-finding trial in multiple solid tumor types that are refractory to standard curative or palliative therapies. The primary endpoint of the Phase 2a is to establish the /recommended Phase 2 Dose (RPTD) of NKTR-102 by measuring the frequency of Dose Limiting Toxicity (DLT). The Phase 2b portion is an open-label, randomized, two-arm study in patients with second-line metastatic colorectal cancer and study participants will be randomized (1:1) to receive either NKTR-102 and cetuximab or irinotecan and cetuximab. The primary endpoint of the Phase 2b portion of the trial is progression-free survival. Secondary endpoints for both the Phase 2a and 2b portion include response rate, response duration, overall survival, standard pharmacokinetics, and incidence of toxicities, including diarrhea and neutropenia.

DETAILED DESCRIPTION:
The Phase 2a portion of this study is completed. The following entries reflect the Phase 2a portion of this study only. The Phase 2b portion of the study was not enrolled. Based on emerging data regarding the corresponding low efficacy of cetuximab in patients with KRAS mutations, as well as revised NKTR-102 clinical development plans, the Phase 2b portion of the study was not completed.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female patients with an ECOG performance score <3 who have any type of solid tumor refractory to standard therapy and who have adequate bone marrow and organ function at screening.

Exclusion Criteria:

* Patients must not have used any CYP3A4 inducers or inhibitors with 2 weeks prior to the first day of study drug treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (4):
- United States (4):
  - Investigator Site - Scottsdale, Scottsdale, Arizona
  - Investigator Site - Louisville, Louisville, Kentucky
  - Investigator Site - Dallas, Dallas, Texas
  - Investigator Site - Tyler, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NKTR-102 100 mg/m2 + Cetuximab | NKTR-102 125 mg/m2 + Cetuximab
Started | 12 | 6
Completed Cycle 1 | 12 | 6
Completed | 0 | 0
Not Completed | 12 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Brain metastases | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Withdrawal of consent | 0 | 1
Not completed — Disease progression | 8 | 3
Not completed — Tx delayed >2 wks, hospitalized for AE | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- NKTR-102 100 mg/m2 + Cetuximab; NKTR-102 125 mg/m2 + Cetuximab: All patients received NKTR-102 in combination with cetuximab. NKTR-102 was administered intravenously (IV) once every 3 weeks (q3w) over 90 minutes on Day 1. Patients were to be enrolled in one of the following sequential dosing cohorts of NKTR-102: 100, 125, 150, or 175 mg/m2. Only the 100 and 125 mg/m2 were enrolled.
- Total: Total of all reporting groups
Arm/Group | NKTR-102 100 mg/m2 + Cetuximab | NKTR-102 125 mg/m2 + Cetuximab | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (16.8) | 65.0 (3.6) | 57.1 (14.9)
Age, Continuous [Median (Full Range); unit: years] | 52.0 [25 to 80] | 65.5 [59 to 70] | 64.0 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 5 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Copies of UGT1A1*28 [Count of Participants; unit: Participants]
  Not detected | 7 | 1 | 8
  One Copy (Heterozygous) | 5 | 4 | 9
  Two Copies (Homozygous) | 0 | 1 | 1
ECOG Performance [Count of Participants; unit: Participants] — GRADE - ECOG PERFORMANCE STATUS
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 4 | 0 | 4
    1 | 8 | 6 | 14
    2 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities
Description: Number of patients with Dose Limiting Toxicities
Time Frame: 12 months
Population: ITT/Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Total: NKTR-102 Overall Total
  All patients received NKTR-102 in combination with cetuximab. NKTR-102 was administered intravenously (IV) once every 3 weeks (q3w) over 90 minutes on Day 1. Patients were to be enrolled in one of the following sequential dosing cohorts of NKTR-102: 100, 125, 150, or 175 mg/m2. Only the 100 and 125 mg/m2 were enrolled.
Arm/Group | NKTR-102 100 mg/m2 + Cetuximab | NKTR-102 125 mg/m2 + Cetuximab | Total
Number analyzed (Participants) | 12 | 6 | 18
Participants
  Dehydration | 0 | 1 | 1
  Diarrhoea | 1 | 1 | 2
  Renal Failure Acute | 0 | 1 | 1

2. Secondary Outcome: Number of Patients With Dose Limiting Toxicities by NCI-CTCAE
Description: Number of patients with Dose Limiting Toxicities by NCI-CTCAE
Time Frame: 12 months
Population: ITT/Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-102 100 mg/m2 + Cetuximab | NKTR-102 125 mg/m2 + Cetuximab | Total
Number analyzed (Participants) | 12 | 6 | 18
Participants
  Dehydration : Any grade | 0 | 1 | 1
  Dehydration : Grade 3 | 0 | 1 | 1
  Diarrhoea : Any grade | 1 | 1 | 2
  Diarrhoea : Grade 3 | 1 | 1 | 2
  Renal Failure Acute : Any grade | 0 | 1 | 1
  Renal Failure Acute : Grade 4 | 0 | 1 | 1

3. Secondary Outcome: Number of Patients With Overall Response
Description: Complete Response is defined as the disappearance of all target lesions. Partial Response is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. The best overall response was the best response recorded from the start of the study drug until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: 12 months
Population: ITT/Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-102 100 mg/m2 + Cetuximab | NKTR-102 125 mg/m2 + Cetuximab | Total
Number analyzed (Participants) | 12 | 6 | 18
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 3 | 0 | 3
  Stable Disease | 2 | 3 | 5
  Progressive Disease | 7 | 1 | 8

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Total: NKTR-102 Overall Tota
  All patients received NKTR-102 in combination with cetuximab. NKTR-102 was administered intravenously (IV) once every 3 weeks (q3w) over 90 minutes on Day 1. Patients were to be enrolled in one of the following sequential dosing cohorts of NKTR-102: 100, 125, 150, or 175 mg/m2. Only the 100 and 125 mg/m2 were enrolled.l
Arm/Group | NKTR-102 100 mg/m2 + Cetuximab | NKTR-102 125 mg/m2 + Cetuximab | Total
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/6 | 1/18
Serious Adverse Events (participants affected / at risk) | 5/12 | 3/6 | 8/18
Other Adverse Events (participants affected / at risk) | 12/12 | 6/6 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-102 100 mg/m2 + Cetuximab (N=12) | NKTR-102 125 mg/m2 + Cetuximab (N=6) | Total (N=18)
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Renal acute failure (Renal and urinary disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-102 100 mg/m2 + Cetuximab (N=12) | NKTR-102 125 mg/m2 + Cetuximab (N=6) | Total (N=18)
Nausea (Gastrointestinal disorders) | 9 | 6 | 15
Diarrhoea (Gastrointestinal disorders) | 9 | 5 | 14
Fatigue (General disorders) | 9 | 3 | 12
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 | 3 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 3 | 11
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 2 | 0 | 2
Vitreous floaters (Eye disorders) | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 5 | 10
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 8
Constipation (Gastrointestinal disorders) | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 5 | 1 | 6
Chills (General disorders) | 3 | 2 | 5
Asthenia (General disorders) | 1 | 2 | 3
Adverse drug reaction (General disorders) | 1 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 1
Skin candida (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0 | 2
Weight decreased (Investigations) | 0 | 2 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 5 | 11
Anorexia (Metabolism and nutrition disorders) | 4 | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 3
Headache (Nervous system disorders) | 2 | 1 | 3
Burning sensation (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 1 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Sinus operation (Surgical and medical procedures) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.